CLINICAL TRIAL: NCT05352295
Title: Evaluation of the Effects of Covid 19 Infection on Bone Remodeling and Bone Fragility
Acronym: CovidBone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: CovidBone
Record Dates: First submitted 2022-01-12; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Bone Remodeling Bone Fragility Resulting From Covid19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- infected: 40 patients admitted to the IRCCS Galeazzi Orthopedic Institute for fracture with Covid 19 infection ascertained by nasal pharyngeal swab during the patients' clinical routine
- not infected ( control): 40 patients admitted to the IRCCS Galeazzi Orthopedic Institute for fracture without Covid 19 infection ascertained by nasal pharyngeal swab during the patients' clinical routine

SUMMARY:
Although SARS-CoV-2 infection and subsequent COVID-19 disease is regarded as a disease that primarily affects the lungs, it can also damage many other organs. This organ damage may increase the risk of long-term health problems, but much remains to be elucidated as to how COVID-19 infection will affect those who have contracted the infection over time. Since SARS-CoV-2 infection mainly affects elderly people, one of the aspects to be evaluated in the near future is its interaction with bone metabolism, which progressively worsens with advancing age. So far, data on bone metabolism in SARS-COV-2 infection are very scarce. Furthermore, it is not clear whether the incidence of osteoporosis and the risk of fracture may increase in patients after recovery from the infection, due to the interaction of their risk factors (old age, smoking, long-term bed rest). term, hypovitaminosis D and steroid treatment) with the COVID-19 inflammatory process. In patients after recovery from severe acute respiratory syndrome (SARS), osteonecrosis and bone abnormalities with reduced bone density were observed, which were partly but not entirely explained by short-term use of steroids. Infections, trauma and injuries induce the production of endogenous signaling mediators of the inflammatory response. Significantly higher serum concentrations of pro and anti-inflammatory cytokines, including IL-6, TNF-α, and IL-10, characterized by severe versus moderate cases, suggest that disease severity may be associated with a "cytokine storm. "[14]. The interaction between inflammatory molecules, such as cytokines, and the bone system is defined as "osteoimmunology" and osteoimmunological mediators, such as RANKL, OPG, RAGE, play a fundamental role in osteoclastogenesis in physiological and pathological conditions. Although the long-term effects of COVID-19 are still unknown, the alleged consequences of the disease would likely be similar to those of coronavirus-related diseases, including SARS (Severe acute respiratory syndrome). In the case of SARS, viral infection-mediated effects have been described that stimulate osteoclatogenesis. Similarly, the current SARS-Cov-2 could have a dual effect, both direct and indirect, on osteoclastogenesis and, consequently, on bone resorption: indirectly by inducing the cytokine storm that promotes bone resorption, direct by stimulating differentiation and osteoclastic activation through the activation of osteoimmunological mediators.

DETAILED DESCRIPTION:
The biological markers under study ( RANKL, OPG, RAGE) will be determined:

- The determinations will be performed on blood samples performed as part of the checks conducted in the normal diagnostic flow and using the residual material not used for routine diagnostics.

Clinical investigations of bone fragility:

* Radiographic investigations performed routinely (pre-operative and immediate post-operative)
* Laboratory tests required by clinical routine:

  * Pre-operative: blood count, coagulation
  * First post-operative sampling (1 post-operative day): complete blood count, coagulation
  * Second post-operative sampling, if performed (3 postoperative day +/- 1 day): blood count and coagulation or each evaluated parameter, the following will be calculated:
* descriptive statistics (mean, standard deviation for variables with normal distribution, median and range for variables not normally distributed)
* differences between the two populations (Covid19 positive and Covid19 negative) by means of parametric or non-parametric tests based on the normality of the distribution of values
* sensitivity, specificity positive and negative predictive values, likelihood ratio for each test and for a combination of them Statistical analyzes will be performed using the GraphPad Prism V.5.03 computer package for Windows (GraphPad Software, San Diego, CA, www.graphpad.com).

ELIGIBILITY:
Inclusion Criteria:

age greater than or equal to 50 years

* patients in the emergency room for fracture of the proximal femur
* subjects of both sexes
* pathologies related to bone fragility (osteoporosis, fractures, parathyroid pathologies).
* signature of the informed consent
* having performed the nasopharyngeal swab for clinical practice to check for SARS Cov2 infection

Exclusion Criteria:

* previous conditions of hypovitaminosis D
* steroid therapy
* Presence of autoimmune diseases or that can create alterations in the inflammatory response

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 80 samples of patients from the IRCCS Galeazzi Orthopedic Institute for fracture, divided into two groups:
  * 40 with Covid 19 infection confirmed by nasal pharyngeal swab in the course of patients' clinical routine
  * 40 without Covid 19 infection confirmed by nasal pharyngeal swab in the course of patients' clinical routine
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
RANKL/OPG ratio difference in Covid infected patients | Pre-operative: CBC, coagulation or First post-operative collection (1 post-operative day): CBC, coagulation or Second post-operative collection, if performed (3 postoperative day +/- 1 day): CBC and coagulation
  Evaluation of any alteration in bone remodeling and increase in bone fragility resulting from Covid19 infection evaluated by means of the RANKL / OPG ratio, an osteoimmunological indicator of bone fragility, measured pre-operative and in the third postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Peretti, MD PhD, Principal Investigator — I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No